CLINICAL TRIAL: NCT04460248
Title: The Efficacy and Safety of Zanubrutinib, Lenalidomide and Rituximab (ZR2) Regimen in Elderly Treatment-naive Patients With Diffuse Large B-cell Lymphoma (DLBCL)
Brief Title: Zanubrutinib, Lenalidomide and Rituximab (ZR2) in Elderly Treatment-naive Patients With Diffuse Large B-cell Lymphoma (DLBCL)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, First Deputy Director of Shanghai Institute of Hematology, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZR2
Record Dates: First submitted 2020-06-25; First posted 2020-07-07 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — zanubrutinib; Lenalidomide; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Zanubrutinib, Lenalidomide and Rituximab (ZR2) (Experimental)
  Interventions: Drug: Zanubrutinib, Lenalidomide and Rituximab (ZR2)

INTERVENTIONS:
Drug: Zanubrutinib, Lenalidomide and Rituximab (ZR2) — Induction therapy:
  The ZR2 regimen will be given from day 1 of each cycle of treatment. Each cycle will last for 21 days. Participants will receive a total of 6 cycles.
  Dosage:
  1. Zanubrutinib, 160 mg bid, po, day 1-21;
  2. Lenalidomide, 25 mg qd, po, day 2-11;
  3. Rituximab, 375 mg/m2, ivgtt, day 1.
  Maintenance therapy:
  Patients who receive complete response or partial response after induction therapy will receive lenalidomide 25 mg qd po during 1-10 days in every 21 days, for a maximum of 2 years.

SUMMARY:
This is a prospective, single-center, open-label, single-arm clinical study designed to evaluate the efficacy and safety of the Zanubrutinib, Lenalidomide and Rituximab (ZR2) regimen in elderly treatment-naive patient with diffuse large B-cell lymphomas.

ELIGIBILITY:
Inclusion Criteria:

* Treatment-naive pathologically confirmed patients with diffuse large B-cell lymphoma (DLBCL)
* Refuse to undergo systemic chemotherapy or not suitable for chemotherapy
* Radiography detects measurable lesions defined as at least 1 clearly defined lesion/nodule with both long and short diameters longer than or equal to 1.5cm
* Life expectancy of at least 3 months determined by researchers
* The patient or his or her legal representative must provide written informed consent prior to any special examination or procedure for the research
* Research drugs have not been used before

Exclusion Criteria:

* The patient has received systemic or local anti-tumor treatment, including chemotherapy, within three weeks before enrollment
* The patient has complications of uncontrolled cardiovascular diseases, blood clotting disorders, connective tissue diseases, serious infectious diseases and other diseases
* Laboratory measures meet the following criteria at screening (unless caused by lymphoma):

  1. Neutrophils<1.5 x 10^9/L
  2. Platelets<80 x 10^9/L
  3. ALT or AST is 2 times higher than the normal upper limit, AKP and bilirubin are 1.5 times higher than normal upper limit
  4. Creatinine is 1.5 times higher than the normal upper limit
* Other concurrent and uncontrolled medical conditions that the researchers believe that they will affect the patient's participation in the study, including patients with psychosis or other known or suspected patients who cannot fully comply with the research protocol
* HIV-infected patients
* Patients with HbsAg positive are required to have negative HBV DNA before entering the group. In addition, if the patient is HBsAg negative but HBcAb positive (regardless of HBsAb status), HBV DNA test is also required, and if the result is positive, anti-viral treatment is also required, and negative HBV DNA is required before entering the group
* Other medical conditions determined by the researchers that may affect the study

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-08-26 (Actual); Primary Completion 2022-02-16 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Complete response rate | At the end of Cycle 6 (each cycle is 21 days)

SECONDARY OUTCOMES:
2-year progression-free survival | 2 years after enrollment
2-year overall survival | 2 years after enrollment
Incidence rate of adverse events | From enrollment to study completion, a maximum of 3 years.

OTHER OUTCOMES:
Single-cell ribonucleic acid (scRNA) sequencing | From enrollment to study completion, a maximum of 3 years.
  scRNA sequencing in tumor tissue

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu PP, Zhu Y, Shi ZY, Wang L, Cheng S, Qian Y, Zhao Y, He Y, Yi HM, Ou-Yang BS, Jiang XF, Li B, Song Q, Mu RJ, Zhao WL. A phase 2 study of zanubrutinib in combination with rituximab and lenalidomide in de novo diffuse large B-cell lymphoma. Blood. 2025 Nov 20;146(21):2561-2573. doi: 10.1182/blood.2025028649. PMID 40829156